CLINICAL TRIAL: NCT01034553
Title: Phase I/II Study of Combination of Aurora Kinase Inhibitor MLN8237 and Bortezomib in Relapsed or Refractory Multiple Myeloma
Brief Title: Aurora A Kinase Inhibitor MLN8237 and Bortezomib in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC088A; NCI-2009-01475 (Registry Identifier: NCI-CTRP); 08-006317 (Other: Mayo Clinic IRB); X14003 (Other: MPI Protocol); MC088A (Other: Mayo Clinic Cancer Center)
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Results first posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-02

CONDITIONS: Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — MLN 8237; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral aurora A kinase inhibitor MLN8237 once daily on days 1-14 and bortezomib IV on days 1, 4, 8 and 11.
  Interventions: Drug: Aurora A kinase inhibitor MLN8237; Drug: bortezomib

INTERVENTIONS:
Drug: Aurora A kinase inhibitor MLN8237 — Given orally
  Other Names: MLN8237
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; PS-341; VELCADE

SUMMARY:
RATIONALE: Aurora A kinase inhibitor MLN8237 and bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I/II trial is studying the side effects and best dose of giving aurora A kinase inhibitor MLN8237 together with bortezomib and to see how well they work in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated doses (MTD) with the combination of MLN8237 and bortezomib. (Phase I) II. To describe the toxicities associated with the combination of MLN8237 and bortezomib. (Phase I) III. To evaluate the overall response rate to the combination of MLN8237 and bortezomib in patients with relapsed or refractory multiple myeloma. (Phase II)

SECONDARY OBJECTIVE:

I. To assess progression-free survival in patients treated with this combination. (Phase II)

II. To assess overall survival in patients treated with this combination.(Phase II)

OUTLINE: This is a phase I dose escalation study followed by a phase II study. Patients receive oral aurora kinase inhibitor MLN8237 once daily on days 1-14 and bortezomib IV on days 1, 4, 8 and 11. Treatment repeats every 28 days for up to 10 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment all patients are followed every 2 months for 1 year and then every 3 months for 1 year.

ELIGIBILITY:
Inclusion

* ANC >= 1500/uL
* AST =< 2.5 x ULN
* Creatinine =< 1.5 x ULN
* Creatinine clearance as calculated by the method of Cockroft and Gault >= 30 mL/minute
* Patients with relapsed or refractory multiple myeloma requiring treatment
* Patients who have received prior bortezomib therapy will be allowed on trial as long as they did not progress during bortezomib or =< 60 days of therapy discontinuation
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential (WOCBP) only (a WOCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months)
* Willingness to return to enrolling institution for follow-up
* Life expectancy >= 12 weeks
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study
* Male subject agrees to use an acceptable method for contraception for the duration of the study
* Patients have a baseline LVEF >= 45% at baseline
* Bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* PLT >= 100,000/uL
* Total bilirubin =<1.5 x upper limit of normal (ULN) or if total bilirubin is > 1.5 x ULN, the direct bilirubin must be =< 2.0 mg/dL
* Measurable disease of multiple myeloma as defined by at least ONE of the following:
* Serum monoclonal protein >= 1.0 g/dL, >= 200 mg of monoclonal protein in the urine on 24 hour electrophoresis, serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio, monoclonal bone marrow plasmacytosis >= 30% (evaluable disease), or measurable plasmacytoma
* ECOG Performance Status (PS) 0, 1, or 2
* Hgb >= 9 g/dl

Exclusion

* Major surgery, open biopsy (excluding bone marrow) or significant traumatic injury =< 4 weeks prior to registration
* Melphalan or other myelosuppressive agents including lenalidomide and non-myelosuppressive agents such as thalidomide or high dose corticosteroids =< 2 weeks prior to registration
* Concurrent use of corticosteroids, but patients may be on chronic steroids (maximum dose 20 mg/day prednisone equivalent) if they are being given for disorders other than myeloma, i.e., adrenal insufficiency, rheumatoid arthritis, etc
* Uncontrolled infection
* Pregnant women or women of reproductive ability who are unwilling to use effective contraception
* Nursing women
* Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 4 weeks after stopping treatment
* Other co-morbidity or psychiatric illness which would interfere with patient's ability to participate in this trial
* Recent history of myocardial infarction in the six months prior to registration
* Uncontrolled angina or electrocardiographic evidence of acute ischemia
* Severe uncontrolled ventricular arrhythmias or electrocardiographic evidence of active conduction system abnormalities
* Cardiac amyloidosis with hypotension (systolic BP less than 100mmHg)
* MGUS or smoldering myeloma
* Serious non-healing wound, or ulcer
* Known hypersensitivity to Bortezomib, boron or mannitol
* Patient has >=Grade 2 peripheral neuropathy within 14 days before enrollment
* Patient has received other investigational drugs with 14 days before enrollment
* Diagnosed or treated for another malignancy within 2 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
* Infection requiring systemic antibiotic therapy within 14 days preceding the first dose of study drug, or other severe infection
* Inability to swallow orally administered medication
* Prior allogeneic bone marrow or organ transplantation
* Patients who are currently receiving digoxin, cyclosporine, tacrolimus or sirolimus
* Severe cardiac comorbidity
* Known positive for HIV or active infectious hepatitis, type A, B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-02; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander K. Stewart, M.D., Study Chair — Mayo Clinic; Shaji K. Kumar, M.D., Principal Investigator — Mayo Clinic
Locations (6):
- United States (6):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of California, San Francisco, San Francisco, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Ohio State University, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I, Dose 0**: Patients receive 25mg aurora A kinase inhibitor MLN8237 once daily on days 1-14 and 1.3mg Bortezomib on days 1, 4,8, and 11.
  Aurora A kinase inhibitor MLN8237: Given orally bortezomib: Given IV
- Phase I, Dose 0: Patients receive 20mg aurora A kinase inhibitor MLN8237 twice daily on days 1-7 and 1.5mg Bortezomib on days 1, 8,15, and 22.
  Aurora A kinase inhibitor MLN8237: Given orally bortezomib: Given IV
- Phase I, Dose 1: Patients receive 30mg aurora A kinase inhibitor MLN8237 twice daily on days 1-7 and 1.5mg Bortezomib on days 1, 8,15, and 22.
  Aurora A kinase inhibitor MLN8237: Given orally bortezomib: Given IV
- Phase I, Dose 2: Patients receive 40mg aurora A kinase inhibitor MLN8237 twice daily on days 1-7 and 1.5mg Bortezomib on days 1, 8,15, and 22.
  Aurora A kinase inhibitor MLN8237: Given orally bortezomib: Given IV
- Phase I, Dose 3: Patients receive 50mg aurora A kinase inhibitor MLN8237 twice daily on days 1-7 and 1.5mg Bortezomib on days 1, 8,15, and 22.
  Aurora A kinase inhibitor MLN8237: Given orally bortezomib: Given IV
- Phase II, Dose 3: Patients receive 50mg aurora A kinase inhibitor MLN8237 twice daily on days 1-7 and 1.5mg Bortezomib on days 1, 8,15, and 22.
  >
  > Aurora A kinase inhibitor MLN8237: Given orally
  >
  > bortezomib: Given IV
Period: Overall Study
Arm/Group | Phase I, Dose 0** | Phase I, Dose 0 | Phase I, Dose 1 | Phase I, Dose 2 | Phase I, Dose 3 | Phase II, Dose 3
Started | 3 | 4 | 3 | 3 | 6 | 7
Completed | 3 | 4 | 3 | 3 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients: All Patients that received oral aurora A kinase inhibitor MLN8237 and bortezomib IV are summarized in this section.
  Aurora A kinase inhibitor MLN8237: Given orally
Arm/Group | All Patients
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 64.5 [46 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 26
Previous treatment [Number; unit: participants] — Previous treatment for this study is defined as any prior therapy given to the patient for treatment of Myeloma.
  participants | 26

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicity (DLT) (Phase I)
Description: Patients were evaluated over the first cycle of treatment for Dose Limiting Toxicities. For this trail DLTs are as follows:
  An AE attributed (definitely, probably, or possibly) to study treatment during cycle 1 and the following criteria:
  Grade 4 Neutropenia Grade 4 Thrombocytopenia, or grade 3 with bleeding Febrile neutropenia Creatinine serum great than 2 times baseline or upper limit of normal Grade 3 or higher Fatigue Grade 3 or higher nausea, vomiting, or diarrhea Any grade 3 or higher Non-hematologic toxicity per NCI CTCAE V4.0 Inability to initiate the scheduled cycle 2, day 1 due to toxicity
  The maximum tolerated dose level (MTD) will be defined as the highest safely tolerated dose.
Time Frame: 28 days
Measure: Number; unit: participants
Groups:
- Dose 0**: Patients receive 25mg aurora A kinase inhibitor MLN8237 once daily on days 1-14 and 1.3mg Bortezomib on days 1, 4,8, and 11.
  >
  > Aurora A kinase inhibitor MLN8237: Given orally
  >
  > bortezomib: Given IV
- Dose 0: Patients receive 20mg aurora A kinase inhibitor MLN8237 twice daily on days 1-7 and 1.5mg Bortezomib on days 1, 8,15, and 22.
  >
  > Aurora A kinase inhibitor MLN8237: Given orally
  >
  > bortezomib: Given IV
- Dose 1: Patients receive 30mg aurora A kinase inhibitor MLN8237 twice daily on days 1-7 and 1.5mg Bortezomib on days 1, 8,15, and 22.
  >
  > Aurora A kinase inhibitor MLN8237: Given orally
  >
  > bortezomib: Given IV
- Dose 2: Patients receive 40mg aurora A kinase inhibitor MLN8237 twice daily on days 1-7 and 1.5mg Bortezomib on days 1, 8,15, and 22.
  >
  > Aurora A kinase inhibitor MLN8237: Given orally
  >
  > bortezomib: Given IV
- Dose 3: Patients receive 50mg aurora A kinase inhibitor MLN8237 twice daily on days 1-7 and 1.5mg Bortezomib on days 1, 8,15, and 22.
  >
  > Aurora A kinase inhibitor MLN8237: Given orally
  >
  > bortezomib: Given IV
Arm/Group | Dose 0** | Dose 0 | Dose 1 | Dose 2 | Dose 3
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 6
participants | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Overall Response Rate to the Combination of MLN8237 and Bortezomib in Patients With Relapsed or Refractory Multiple Myeloma.
Description: sCR: Normal serum FLC ratio, and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence, negative immunofixation of the serum and urine, <5% plasma cells in bone marrow, disappearance of any soft tissue plasmacytomas, and normalization of FLC ratio. VGPR:PR and serum and urine M-component detectable by immunofixation but not on electrophoresis, or if serum measurable,≥90% or greater reduction in serum M-component plus urine M-component <100 mg per 24h and if only measurable non-bone marrow parameter was FLC,≥90% or greater reduction in difference from involved and uninvolved FLC levels. PR:≥50% reduction of serum M-protein or reduction in 24-h urinary M-protein by ≥90% or to <200 mg per 24h or if FLC, ≥50% decrease in the difference between involved and uninvolved FLC levels or ≥50% reduction in bone marrow plasma cells is required in place of M-protein, provided baseline percentage was ≥30%, and ≥50% reduction in the size of soft tissue plasmacytomas
Time Frame: Every 28 day cycle(up to 10 cycles)
Population: All patients that received treatment were evaluated.
Measure: Number; unit: percentage of patients per dose level
Groups:
- Dose Level 0: This includes patients who received 25mg aurora A kinase inhibitor MLN8237 once daily on days 1-14 and 1.3mg Bortezomib on days 1, 4,8, and 11. As well as, patients who received 20mg aurora A kinase inhibitor MLN8237 twice daily on days 1-7 and 1.5mg Bortezomib on days 1, 8,15, and 22.
- Dose Level 1: Patients received 30mg aurora A kinase inhibitor MLN8237 twice daily on days 1-7 and 1.5mg Bortezomib on days 1, 8,15, and 22.
- Dose Level 2: Patients received 40mg aurora A kinase inhibitor MLN8237 twice daily on days 1-7 and 1.5mg Bortezomib on days 1, 8,15, and 22.
- Dose Level 3: Patients received 50mg aurora A kinase inhibitor MLN8237 twice daily on days 1-7 and 1.5mg Bortezomib on days 1, 8,15, and 22.
Arm/Group | Dose Level 0 | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 7 | 3 | 3 | 13
percentage of patients per dose level
  Strong Complete Response | 14.3 | 0 | 0 | 0
  Very Good Partial Response | 0 | 33.3 | 0 | 7.7
  Partial Response | 14.3 | 0 | 0 | 23.1

3. Secondary Outcome: Progression-free Survival
Time Frame: Every 28 day cycle(up to 10 cycles) then follow-up for up to 2 years
Population: All patients that received treatment were evaluated.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- All Patients: Patients receive oral aurora A kinase inhibitor MLN8237 once daily on days 1-14 and bortezomib IV on days 1, 4, 8 and 11.
  >
  > Aurora A kinase inhibitor MLN8237: Given orally
  >
  > bortezomib: Given IV
Arm/Group | All Patients
Number analyzed (Participants) | 26
Months | 5.9 [4.1 to 15.8]

4. Secondary Outcome: Overall Survival
Time Frame: Every 28 day cycle(up to 10 cycles) then follow-up for up to 2 years
Population: All patients that received treatment were evaluated.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- All Patients: Patients receive oral aurora A kinase inhibitor MLN8237 and bortezomib IV. >
  > Aurora A kinase inhibitor MLN8237: Given orally
  >
  > bortezomib: Given IV
Arm/Group | All Patients
Number analyzed (Participants) | 26
Months | 23.6 [17.4 to NA] — Insufficient number of participants with events

ADVERSE EVENTS:
Groups:
- All Patients: bortezomib: Given IV
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 11/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=26)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 3 (5)
Urinary tract infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (4)
Neutrophil count decreased (Investigations) | 5 (11)
Platelet count decreased (Investigations) | 2 (7)
White blood cell decreased (Investigations) | 3 (6)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=26)
Anemia (Blood and lymphatic system disorders) | 10 (24)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 16 (52)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 5 (7)
Nausea (Gastrointestinal disorders) | 18 (79)
Vomiting (Gastrointestinal disorders) | 9 (14)
Edema limbs (General disorders) | 1 (9)
Fatigue (General disorders) | 21 (93)
Fever (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 11 (29)
Lung infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (36)
Creatinine increased (Investigations) | 7 (15)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
INR increased (Investigations) | 1 (5)
Lymphocyte count decreased (Investigations) | 8 (33)
Neutrophil count decreased (Investigations) | 12 (61)
Platelet count decreased (Investigations) | 22 (128)
Weight loss (Investigations) | 3 (3)
White blood cell decreased (Investigations) | 7 (35)
Anorexia (Metabolism and nutrition disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (3)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 7 (46)
Peripheral sensory neuropathy (Nervous system disorders) | 17 (111)
Somnolence (Nervous system disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (24)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (7)
Hypertension (Vascular disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes